CLINICAL TRIAL: NCT01643538
Title: Social Goals and Individual Incentives to Promote Walking in Older Adults (Way to Walk II)
Brief Title: Social Goals and Individual Incentives to Promote Walking in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69924
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-02

CONDITIONS: Physical Activity
Keywords: physical activity; adults age 65 and older; financial incentives
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Arm (Active Comparator): Daily use of pedometer for 5 months. Walking goal set based on level of walking during 2-week run-in period. Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week.
  Subjects in the Control Group will only receive pedometers and weekly feedback on their performance through the same mechanisms and with the same frequency as participants in the other three study arms. There will be no financial incentives or charity donations in this group.
  Interventions: Behavioral: daily pedometer use and weekly feedback
- Personal Financial Incentives Arm (Experimental): Daily use of pedometer for 5 months. Walking goal set based on level of walking during 2-week run-in period. Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week. Each week, if pedometer is used and walking goal is met for 5 out of 7 days, participant will receive $20. Financial incentive is terminated after 4 months. Daily use of pedometer continues for an additional 4 weeks.
  Interventions: Behavioral: Financial incentive; Behavioral: daily pedometer use and weekly feedback
- Social Goals Arm (Experimental): Daily use of pedometer for 5 months. Walking goal set based on level of walking during 2-week run-in period. Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week. Each week participants will be asked to designate which charity should receive a donation if they meet or exceed their goal. If they meet the goal, they will be notified that a donation of $20 in their name has been sent to the charity. Charity donation is terminated after 4 months. Daily use of pedometer continues for an additional 4 weeks.
  Interventions: Behavioral: Social Goal; Behavioral: daily pedometer use and weekly feedback
- Combined Financial Incentives & Social Goals Arm (Experimental): Daily use of pedometer for 5 months. Walking goal set based on level of walking during 2-week run-in period. Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week. Each week, the participant will be asked to choose whether to keep, give, or split the reward, if they meet or exceed their goal. If they choose to send some of the money to charity, they will be asked to identify a charity to which they would like to donate the payment. If they meet their goal, they will receive money and/or be notified that a donation of the selected amount has been sent to the charity, depending on their selected preference. Incentives are terminated after 4 months. Daily use of pedometer continues for an additional 4 weeks.
  Interventions: Behavioral: Personal financial incentives & social goals; Behavioral: daily pedometer use and weekly feedback

INTERVENTIONS:
Behavioral: Financial incentive — Participants will receive a direct financial incentive in the amount of $20 for each week when their daily pedometer step count equals or exceeds their goal at least 5 out of 7 days.
  Arms: Personal Financial Incentives Arm
Behavioral: Social Goal — Participants will be asked to identify a charity to which they would like to donate the payment for reaching their walking goal. Each week they will be asked to designate which charity should receive a donation if they meet or exceed their goal. If they meet the goal, they will be notified that a donation of $20 in their name has been sent to the charity.
  Arms: Social Goals Arm
Behavioral: Personal financial incentives & social goals — Participants will be able to allocate their reward for reaching their walking goal: the $20 reward can be divided between personal financial incentive and a charitable donation. Each week, the participant will be asked to choose whether to keep, give, or split the reward, if they meet or exceed their goal. If they choose to send some of the money to charity, they will be asked to identify a charity to which they would like to donate the payment. If they meet their goal, they will be notified by email or mail (based on their preference), that a donation of the selected amount has been sent to the charity.
  Arms: Combined Financial Incentives & Social Goals Arm
Behavioral: daily pedometer use and weekly feedback — Daily use of pedometer for 5 months. Walking goal set based on level of walking during 2-week run-in period. Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week.

SUMMARY:
The goal of this randomized and controlled trial is to test whether a financial incentive of a donation to achieve a social goal is more effective to motivate and sustain a daily walking habit than the same dollar value given to an older adult. The investigators will achieve this using a novel computer platform utilizing a digital pedometer-internet interface.

ELIGIBILITY:
Inclusion Criteria:

* Adult 65 years of age and older
* Can read and speak English
* Access to a personal computer with high-speed internet connection and functional Universal Serial Bus (USB) port for the study duration
* Able to walk 1/4 mile (i.e., 2 to 3 blocks) without stopping
* No pedometer use in last 30 days

Exclusion Criteria:

Major medical conditions including:

* serious heart and lung diseases
* diabetes requiring insulin therapy
* severe arthritis
* neurologic disorders
* dementia
* heavy alcohol use
* recent knee or spinal surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
mean proportion of days that step per day goals were attained | 16 weeks

SECONDARY OUTCOMES:
mean number of steps per day | 16 weeks
mean proportion of days that step per day goals were attained during follow-up | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — University of Pennsylvania; Jason Karlawish, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Harkins KA, Kullgren JT, Bellamy SL, Karlawish J, Glanz K. A Trial of Financial and Social Incentives to Increase Older Adults' Walking. Am J Prev Med. 2017 May;52(5):e123-e130. doi: 10.1016/j.amepre.2016.11.011. Epub 2017 Jan 3. PMID 28062271